CLINICAL TRIAL: NCT02770235
Title: Evaluation of Advanced Glycation End-products (AGE) and the Erectile Dysfunction (DE) in Diabetic Patients
Acronym: APGADEPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PI2013_843_0021
Record Dates: First submitted 2016-05-11; First posted 2016-05-12 (Estimated); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Diabetes Mellitus, Non-Insulin-Dependent; Erectile Dysfunction
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Erectile Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DE assessment and AGE measurements (Experimental): To evaluate the association between erectile dysfunction (DE) and AGE levels by using non-invasive measurement AGE-ReaderTM, in diabetic patients
  Interventions: Other: DE assessment; Other: AGE measurement

INTERVENTIONS:
Other: DE assessment — by a validated self-administered questionnaire: Index International erectile function (IIEF-15)
Other: AGE measurement — By AGE-ReaderTM

SUMMARY:
In diabetics there is an abnormally increased production of AGEs due to hyperglycemia. An association was shown between AGE measured by biopsy (invasive) and DE patients with diabetes (increase of AGE level in the corpora cavernosa). To date no studies have explored the link between DE and the measure of AGE by a non-invasive method of Auto-fluorescence (AF) Skin (AGEReaderTM).

If the hypothesis of an association between DE and AGE measured by AF was checked, screening for erectile dysfunction and measurement of AGEs could help to improve the overall management of diabetic patient (including cardiovascular) and their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes Type 2

Exclusion Criteria:

* skin hyperpigmentation

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2014-03-17 (Actual); Primary Completion 2019-03-16 (Actual); Study Completion 2019-03-16 (Actual)

PRIMARY OUTCOMES:
erectile dysfunction and AGE levels | 2 hours
  To evaluate the association between erectile dysfunction and AGE levels by using non-invasive measurement AGE-ReaderTM, in diabetic patients

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Daniel LALAU, MD PhD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France

REFERENCES:
- [Result] Kouidrat Y, Zaitouni A, Amad A, Diouf M, Desailloud R, Loas G, Lalau JD. Skin autofluorescence (a marker for advanced glycation end products) and erectile dysfunction in diabetes. J Diabetes Complications. 2017 Jan;31(1):108-113. doi: 10.1016/j.jdiacomp.2016.10.026. Epub 2016 Oct 29. PMID 27847146